CLINICAL TRIAL: NCT00065975
Title: Physical CAM Therapies for Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AT000622-01 (NIH); EisenbergD
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; acupuncture; chiropractic; massage therapy; CAM therapies
MeSH Terms: interventions — Massage; Manipulation, Chiropractic; Acupuncture Therapy

INTERVENTIONS:
Procedure: massage therapy
Procedure: chiropractic
Procedure: acupuncture

SUMMARY:
This is a pilot randomized trial intended to evaluate the effectiveness of acupuncture, chiropractic and massage for chronic back pain in older and younger adults.

ELIGIBILITY:
* Low back pain duration of at least 3 months;
* Low back pain occurring in the past week;
* No numbness or tingling in the lower extremities;
* No pain that radiates to below the knee;
* No use of massage, chiropractic or acupuncture for any reason in the past year;
* Able to attend scheduled appointments;
* Able to hear, read, and understand English;
* No low back pain surgery in the past 3 years;
* No unexplained weight loss;
* No previous vertebral or spinal fractures;
* No previous non-traumatic bone fractures;
* No other spinal pathology, including scoliosis, spinal stenosis, osteoporosis, or ankylosing spondylitis;
* No cancer (except simple skin cancers) in the past 5 years;
* No pacemakers;
* No bleeding problems or anticoagulant use;
* No major organ transplants;
* No oral corticosteroid use for more than 4 consecutive weeks during the past year;
* Cannot be pregnant;
* Must be able to get down to and up from the floor by yourself;
* Able to walk 2 flat city blocks unassisted;
* Willing to participate in periodic telephone interviews.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-04; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: David Eisenberg, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (2):
- United States (2):
  - Harvard medical school, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Boston, Massachusetts